CLINICAL TRIAL: NCT05419583
Title: Targeting Investigation and Treatment in Patients With Type 2 Myocardial Infarction (TARGET-Type 2): A Pilot Randomised Controlled Trial
Brief Title: Targeting Investigation and Treatment in Patients With Type 2 Myocardial Infarction
Acronym: TARGET-Type 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC22023
Record Dates: First submitted 2022-06-03; First posted 2022-06-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Myocardial Infarction Type 2
Keywords: Type 2 myocardial infarction; Randomised controlled trial; Fourth Universal Definition of Myocardial Infarction; Coronary artery disease; Left ventricular systolic dysfunction
MeSH Terms: conditions — Coronary Artery Disease; Ventricular Dysfunction, Left | interventions — Echocardiography; Platelet Aggregation Inhibitors; Aspirin; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Anticoagulants; apixaban; edoxaban; Warfarin; Cardiovascular Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Patients will continue to be treated by the clinical team based on NHS guidelines. They will receive no additional visits from the study however may be asked to participate in qualitative interviews at the end of the study about their usual care. The standard care pathway may involve further investigation with clinically indicated tests or treatments and no appropriate tests or treatments will be withheld.
- Complex intervention (Experimental): A structured risk assessment for coronary disease or left ventricular impairment and management plan delivered by a cardiologist to guide targeted investigation and treatment. This may include imaging with coronary computed tomography angiography (CCTA), invasive coronary angiography, transthoracic echocardiography or cardiac MRI. Treatments may include antiplatelet and anticoagulant therapy, statin therapy or treatments for heart failure as indicated in line with international guidelines.
  Interventions: Diagnostic Test: Coronary computed tomography angiography; Diagnostic Test: Invasive coronary angiography; Diagnostic Test: Transthoracic echocardiography; Diagnostic Test: Cardiac MRI scan; Drug: Antiplatelet Drug (Aspirin or Statin); Drug: Anticoagulants (Apixaban, Edoxaban, Rivaroxoban, Warfarin); Drug: Guideline directed heart failure therapy; Drug: Statins (Cardiovascular Agents)

INTERVENTIONS:
Diagnostic Test: Coronary computed tomography angiography — CT scan of the heart arteries
  Arms: Complex intervention
Diagnostic Test: Invasive coronary angiography — Invasive coronary angiography via the radial or femoral approach
  Arms: Complex intervention
Diagnostic Test: Transthoracic echocardiography — Ultrasound scan of the heart
  Arms: Complex intervention
Diagnostic Test: Cardiac MRI scan — An MRI scan to assess the heart structure and function
  Arms: Complex intervention
Drug: Antiplatelet Drug (Aspirin or Statin) — Antiplatelet therapy for coronary artery disease
  Arms: Complex intervention
Drug: Anticoagulants (Apixaban, Edoxaban, Rivaroxoban, Warfarin) — Anticoagulant therapy if atrial fibrillation identified (DOAC or Warfarin)
  Arms: Complex intervention
Drug: Guideline directed heart failure therapy — Use of guideline approved heart failure treatments (ACE-inhibitor / angiotensin receptor blocker (ARB) / ARB and neprilysin inhibitor, mineralocorticoid receptor antagonist, beta blocker, SGLT-2 inhibitor, diuretic therapy)
  Arms: Complex intervention
Drug: Statins (Cardiovascular Agents) — Statins will be recommended for patients with coronary plaque disease or hypercholesterolaemia
  Arms: Complex intervention

SUMMARY:
Type 2 myocardial infarction (MI) is common and associated with poor clinical outcomes, with as many as one in ten experiencing recurrent MI within one year, and only one in three alive at five years. Recent prospective data demonstrates two-thirds of patients with type 2 MI have underlying coronary artery disease and one-third have left ventricular systolic impairment. Importantly, this is previously unrecognised in over half of all patients, suggesting there may be opportunities to identify and treat these underlying conditions to modify clinical outcomes. The investigators will undertake a pilot randomised controlled trial in which patients will be randomised to standard care or a complex intervention involving detailed cardiology assessment for the likelihood of coronary disease or left ventricular impairment, followed by targeted investigation and treatment where underlying disease is identified. This study will inform the design and delivery of a prospective multi-centre randomised controlled trial powered for clinical outcomes.

DETAILED DESCRIPTION:
TARGET-Type 2 is the pilot phase of a prospective, randomised, open label with blinded endpoint evaluation (PROBE) parallel group, event driven, multicentre trial, assessing the impact of a complex intervention in patients hospitalised with type 2 myocardial infarction. Patients will be recruited from the Royal Infirmary of Edinburgh, Edinburgh (tertiary cardiac referral centre) and the Victoria Hospital, Kirkcaldy (district general hospital). The study aims to recruit 60 patients with type 2 myocardial infarction who will be randomised 1:1 to standard care or the complex intervention.

Potential participants will be identified throughout the hospital, including the Emergency Department (ED), Acute Medical Unit (AMU) and all inpatient wards whilst in hospital and using electronic medical records after discharge. Potential participants who are not approached in hospital (e.g., as they attend out of hours or due to the lack of availability of the study team) will be identified using electronic medical records or through referral from the clinical team and contacted by phone by the research team to invite them to take part in the study. The trial will be integrated into routine clinical care at participating sites. A pre-screening log will be kept of patients who meet the inclusion criteria and are subsequently found to be ineligible or not recruited.

Following consent and completion of baseline assessments patients who meet all inclusion/exclusion criteria and are eligible will be randomised into the study, using a web-based computer-generated randomisation process.

Patients will be randomised 1:1 ratio to either standard care or the complex intervention. Randomisation will be stratified based on the presence of 1) known coronary artery disease and 2) known left ventricular systolic dysfunction. Once randomised, a letter will be sent to the participant's General Practitioner (GP) to inform them of their involvement in the study and treatment allocation. Study participants who are randomised to usual care will not have any additional study visits. Those randomised to the complex intervention may be invited for further investigations to guide additional treatment and invited for follow up clinic visits.

Proposed Complex Intervention: A structured management plan for doctors to guide their (a) risk assessment, (b) targeted investigation and (c) secondary preventative therapy delivered after consultation with a cardiologist. All investigations and treatments recommended are established practice in national and international clinical guidelines for patients with coronary artery disease or LV impairment due to type 1 MI.

The cardiologist will estimate if the pre-test probability of coronary artery disease or LV impairment is low, intermediate, or high. This assessment will be based on symptoms, cardiovascular risk factors, previous medical history, and an evaluation of the presenting illness and initial routine investigations including a physical examination, routine blood tests, the 12-lead ECG and chest x-ray.

Where the probability of coronary disease or LV impairment is low, further investigation may not be indicated. Where the probability of coronary artery disease is intermediate, coronary computed tomography angiography (CCTA) may be recommended. CCTA will be performed according to previously published methodology. Patients with a heart rate exceeding 65 beats/min will receive oral beta-blockade (50 or 100 mg metoprolol) 1 hour before computed tomography. Additional intravenous beta blockers will be given depending on heart rate at the time of imaging. All patients will receive sublingual glyceryl trinitrate (300 μg) immediately prior to dual cardiac and respiratory-gated computed tomography imaging of the coronary arteries. The investigators will quantify total plaque burden using CT calcium scoring. A bolus of 80-100 mL of contrast (400 mg/mL; Iomeron, Bracco, Milan, Italy) will be injected intravenously at 5 mL/s. CT angiography will be evaluated jointly by a Radiologist and a Cardiologist with suitable training to determine the extent of coronary atherosclerosis.

In select cases, where the probability of obstructive coronary disease is considered high or if the patient has ongoing symptoms of myocardial ischaemia, invasive coronary angiography may be recommended. Where invasive coronary angiography is recommended this will be performed via the femoral or radial artery with 6F arterial catheters. Where coronary artery disease is known or highly likely, no further investigations may be required unless there is clinical suspicion of worsening disease severity.

Where the probability of LV impairment is intermediate or high, a transthoracic echocardiogram will be recommended. Standard transthoracic echocardiography will be undertaken in accordance with guidance from the British Society of Echocardiography for 'full examination'. In selected patients where there is a suspicion of underlying cardiomyopathy or recent type 1 MI based on abnormal findings on echocardiography, cardiovascular magnetic resonance (CMR) and coronary imaging if not already performed will be considered to identify areas of scar or to clarify the final diagnosis in line with usual recommendations for clinical practice. It is intended that where possible, investigations will be completed within thirty days of randomisation.

The investigators will identify if there is coronary heart disease or left ventricular impairment in patients with type 2 myocardial infarction. Our treatment strategy will involve the use of therapies approved by clinical guidelines for use in standard clinical practice because of proven benefit for the secondary prevention of cardiovascular events in patients with coronary artery disease with anti-platelet agents, such as aspirin or P2Y12 inhibitors, and lipid lowering drugs, such as statins. In patients who undergo invasive coronary angiography, if there is evidence of recent plaque rupture or where there are high risk features, revascularisation with percutaneous coronary intervention will be considered if in the patient's best interests, in line with clinical practice guidelines. Revascularisation will also be considered in patients with obstructive coronary artery disease who report limiting anginal symptoms despite medical therapy. This intervention may be considered at the first procedure where patients are established on treatment, or during follow up review.

In patients with evidence of left ventricular impairment, additional therapies including beta blockers, angiotensin converting enzyme (ACE) or angiotensin receptor blocker (ARB) or aldosterone/neprilysin inhibitors, mineralocorticoid receptor antagonists (MRA) and SGLT-2 inhibitors will be considered and recommended in line with guideline recommendations. All drugs have a class I recommendation from the European Society of Cardiology in patients with left ventricular impairment. Decision making on treatment recommendations will be patient centred, and whilst recommendations will be made by the study team all prescriptions will issued by the usual care team after consideration.

Patients found to have obstructive coronary artery disease, moderate to severe LV impairment, evidence of cardiomyopathy or at least moderate valvular heart disease will be offered a cardiology outpatient clinic appointment for further assessment. A structured template recording a clinical summary, cause of type 2 MI, assessment, investigation and treatment recommendations will be recorded on the electronic patient record for the usual care team. A letter will be sent to the GP informing them of participation in the study, treatment allocation, the results of investigations and recommended treatments. In those who provide consent, blood samples will be obtained to facilitate biomarker evaluation and risk stratification in future studies

As recruitment to the TARGET-Type 2 feasibility study begins, recruitment processes will be investigated using qualitative research methods to identify specific facilitators or barriers to recruitment. a purposive sample of patients across a range of ages, trial participation status and study site will also be invited to consent to an interview study. Interviews will explore reasons for participation and non-participation, and the acceptability of study procedures. Patients can choose whether to take part in either or both parts of the study. Interviews with patients will explore views on the presentation of trial information, understanding of study processes (e.g. randomisation), the acceptability of study interventions and reasons underlying decisions to consent or decline to participate. If screening logs identify clinician hesitation to randomise their patient as a barrier to recruitment, clinicians will be invited to participate in an interview to explore the reasons underpinning this. The interview topic guide will explore views about the trial importance, relevance and interventions from a clinician's point of view, and how recruitment operates in practice.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with a clinical diagnosis of type 2 myocardial infarction, defined as:

i. Symptoms of myocardial ischaemia, or signs of myocardial ischaemia on 12-lead electrocardiogram (≥0.5mm ST segment depression in any two contiguous leads or new regional T wave inversion)

ii. A clinically significant change in high-sensitivity cardiac troponin concentration with at least one value above the 99th centile upper reference limit, or a single measurement if considered significantly elevated

iii. Documented evidence of myocardial oxygen supply (anaemia, hypoxia, hypotension, bradycardia, tachycardia, arrhythmia) or demand (hypertension, left ventricular hypertrophy, valvular heart disease) imbalance.

Exclusion Criteria:

i. Patients under 30 years who are less likely to benefit from cardiac imaging

ii. Inability to give informed consent

iii. Patients on renal replacement therapy or with eGFR <30ml/min

iv. Patients with advanced frailty (based on Clinical Frailty Score ≥7)

v. Patients who are pregnant or breast feeding

vi. Patients with ST-segment elevation on 12-lead electrocardiogram

vii. Patients with a clinical diagnosis of type 1 myocardial infarction

viii. Patients who have had diagnostic imaging confirming coronary vasospasm, embolism or spontaneous coronary artery dissection has caused type 2 myocardial infarction

ix. Previous randomization into TARGET-Type 2 pilot study

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Trial process outcomes: eligibility, approach, consent and randomisation | 90 days
  The proportion of patients who are eligible, approached, consented and randomised

SECONDARY OUTCOMES:
Recruitment rate | 30 days and 90 days
  Rate per month and overall
Adherence to recommended investigation | 90 days
  Determined as the proportion of patients who received recommended investigation
Adherence to recommended treatment | 90 days
  Determined as the proportion of patients who received recommended treatment
Proportion of patients with changes in prescription of secondary prevention therapy | 90 days
  Defined as initiation, intensification or cessation of cardiac medication including aspirin, clopidogrel, statin, bisoprolol or ACE-inhibitor and others as defined in data dictionary.
Frequency of investigation and treatment | 90 days
  Proportion of patients who undergo routine cardiac investigation (echocardiography, invasive coronary angiography, percutaneous coronary intervention, CT coronary angiography, cardiac MRI) in the standard care arm per month
Change in classification of myocardial infarction | 90 days
  Proportion of patients in whom the classification of myocardial infarction changes after study intervention
Quantity of missing data | Baseline and 90 days

OTHER OUTCOMES:
Rate of myocardial infarction | 90 days
  As per the Fourth Universal Definition
Rate of all-cause death | 90 days
Rate of cardiovascular death | 90 days
  Defined as death resulting from an acute myocardial infarction, sudden cardiac death, death due to heart failure, death due to stroke, death due to haemorrhage, and death due to other cardiovascular causes
Rate of cardiac death | 90 days
  Defined as death resulting from an acute myocardial infarction, sudden cardiac death, or death due to heart failure.
Rate of non-cardiovascular death | 90 days
  Defined as death arising from any other cause not listed under cardiovascular death
Rate of hospitalisation with heart failure | 90 days
Rate of unscheduled coronary revascularization | 90 days
Rate of major bleeding | 90 days
  Bleeding Academic Research Consortium [BARC] 3-5

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Chapman, MBChB PhD, Study Chair — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - Victoria Hospital, Kirkcaldy, Fife
  - NHS Lothian, Edinburgh, Lothian

IPD SHARING:
Plan to Share IPD: Undecided
Requests for IPD will be considered on an individual basis in line with ethical and regulatory approvals